CLINICAL TRIAL: NCT03298581
Title: An Open-label Safety Study to Assess the Multiple-dose Pharmacokinetics and Potential for Adrenal Suppression Following Topical Treatment With Halobetasol Propionate 0.05% Topical Spray Applied Twice Daily for 28 Days in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Multiple-Dose Pharmacokinetics and Potential for Adrenal Suppression Following Treatment With Halobetasol Spray in Patients With Plaque Psoriasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 71542610
Record Dates: First submitted 2017-09-19; First posted 2017-10-02 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — halobetasol; Therapeutics

STUDY DESIGN:
Intervention Model Description: Open label, single treatment arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Halobetasol propionate spray 0.05% (Experimental): Patients will instructed o apply halobetasol spray twice daily for 14 days and not to rub over the affected area after application of spray.
  Interventions: Drug: Halobetasol Propionate

INTERVENTIONS:
Drug: Halobetasol Propionate — Experimental: Treatment with topical halobetasol spray 0.05% Patients will instructed o apply halobetasol spray twice daily for 28 days and not to rub over the affected area after application of spray.
  Other Names: Topical treatment with Halobetasol spray

SUMMARY:
This is an open-label, safety study designed to assess the multiple-dose pharmacokinetics and potential for adrenal suppression following topical treatment with halobetasol propionate 0.05% spray applied twice-daily in adult patients with moderate to severe plaque psoriasis. At least 40 eligible patients with plaque psoriasis that satisfy all eligibility criteria will be enrolled into the study

DETAILED DESCRIPTION:
This is an open-label, safety study designed to assess the multiple-dose pharmacokinetics and potential for adrenal suppression following topical treatment with halobetasol propionate 0.05% spray applied twice-daily in adult patients with moderate to severe plaque psoriasis. At least 40 eligible patients with plaque psoriasis that satisfy all eligibility criteria will be enrolled into the study. Patients must be overall in good health and should have a current diagnosis of moderate to severe plaque psoriasis with Investigator Global Assessment (IGA) score of at least 3 or 4. Patients will be stratified by age with:

Cohort 1: At least 20 patients 18 years of age and older with ≥ 20% body surface area (BSA) affected Cohort 2: At least 20 patients 12-16 years and 11 months of age with ≥ 10% BSA affected Cohort 2 will initiate enrollment once all enrolled patients in Cohort 1 have completed the study and a safety analysis has been reviewed by the Medical Monitor and approved by the Novum Independent Institutional Review Board (NIIRB). Sites will not begin enrollment of patients in Cohort 2 until the site is notified by email that the safety analysis for Cohort 1 has been reviewed and approved. Confirmation of email receipt will be required from each Investigator before enrollment of Cohort 2 can begin. Each cohort will be enrolled based on the availability of patients. Each cohort will be reviewed for the potential of HPA axis suppression. The Medical Monitor or NIIRB may discontinue the study at any time if safety concerns are found. If 6 or more patients in Cohort 1 experience HPA axis suppression, then enrollment for Cohort 1 will be stopped. Cohort 2 will not be initiated if 6 or more patients enrolled in Cohort 1 experience HPA axis suppression or 30% or more of the final enrolled number of patients in Cohort 1 experience HPA axis suppression. If 6 or more patients in Cohort 2 experience HPA axis suppression, then enrollment for Cohort 2 will be stopped. If the study is stopped at any time, patients currently enrolled will be contacted via phone and instructed to discontinue study product immediately. Patients will be instructed to return for their next scheduled visit for cortisol response testing. Sites will follow up with patients and monitor for HPA axis suppression. All patients will be followed until cortisol levels are normal.

Patients will be instructed to apply topical spray twice daily onto the affected skin areas for 28 days. Patients will be instructed not to rub over the affected area after application of spray Patients will apply the morning dose of the study product in the clinic at each clinic visit and at home during non-clinic visits. A phone call will be made approximately 14 days after the patient has completed dosing to follow-up on any new adverse events that may have occurred

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females:

   * Cohort 1: 18 years of age and older
   * Cohort 2: 12-16 years and 11 months of age (Cohort 2 will not begin enrollment until review and approval of safety information from Cohort 1.)
2. If female and of childbearing potential, prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom, IUD, oral, transdermal or injected hormonal contraceptives). Female patients using hormonal contraceptives should have been on the same product/dosing regimen for at least 28 days before baseline and should not change this regimen during the study.
3. Signed informed consent form that meets all criteria of current FDA regulations. For a patient considered to be a minor in the state he/she lives and is enrolled, the parent or legal guardian will be required to sign the consent form and the patient will sign an IRB approved "assent to participate" form. Approved informed consent and assent forms specific to each cohort will be required.
4. Patients with a definite clinical diagnosis of stable plaque psoriasis with:

   * Cohort 1: 18 years of age and older with ≥ 20% BSA affected (excluding the face, scalp, groin, axillae and other intertriginous areas)
   * Cohort 2: 12-16 years and 11 months of age with ≥ 10% BSA affected (excluding the face, scalp, groin, axillae and other intertriginous areas)
5. Investigator Global Assessment (IGA) score of 3 (Moderate) or 4 (Severe).
6. Patients in Cohort 2 must weigh a minimum of 24 kg.
7. Results from a cortisol response test that are considered normal and show no evidence of any abnormal HPA function or adrenal response. Patients must fulfill all of the following stipulations:

   1. Basal (pre-Cortrosyn™ injection) cortisol concentration ≥ 5 mcg/100 mL.
   2. 30-minute post-injection cortisol level is at least 7 mcg/100 mL greater than the basal level (≥ basal value + 7).
   3. Post-stimulation level > 18 mcg/100 mL.

Exclusion Criteria:

1. Females who are pregnant, nursing, planning to become pregnant during the duration of the study, or if of childbearing potential and sexually active and not prepared to use appropriate contraceptive methods to avoid pregnancy.
2. Lacks stable diagnosis of plaque psoriasis or has been diagnosed with mild plaque psoriasis.
3. IGA score < 3.
4. Plaque psoriasis with a BSA involvement < 20% for Cohort 1 or < 10% for Cohort 2.
5. Current diagnosis of types of psoriasis other than stable plaque psoriasis (i.e., erythrodermic, exfolative or pustular psoriasis).
6. Results from a cortisol response test that show evidence of any abnormal HPA function or adrenal response:

   1. Basal (pre-CortrosynTM injection) cortisol concentration < 5 mcg/100 mL.
   2. 30-minute post-injection cortisol level is less than 7 mcg/100 mL greater than the basal level (< basal value + 7).
   3. Post-stimulation level ≤ 18 mcg/100 mL.
7. Patient has a history of plaque psoriasis that has been unresponsive to topical corticosteroid therapy.
8. Any condition (i.e., sunburn, atopic or contact dermatitis, etc.) that, in the Investigator's opinion, may interfere with the clinical assessments of the signs and symptoms of plaque psoriasis.
9. History of prolonged bleeding or a past diagnosis of bleeding disorders and/or history of blood loss exceeding 450 mL (including blood donations) within 1 month before the study.
10. Patient with poor peripheral venous access.
11. History of mastectomy or lymphatic insufficiency of the upper limb (patient is eligible if blood can be taken from the arm opposite the site of surgery or condition).
12. History of allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance that in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.
13. Patient has a significant history or current evidence of chronic infectious disease, system disorder, Netherton's Syndrome, uncontrolled diabetes, organ disorder or insufficiency, immunosuppression (from medical treatment or disease) or other medical condition (including active or recurrent bacterial, viral or fungal infection or open wounds) that, in the Investigator's opinion, would place the study patient at undue risk by participation in the study or as an unsuitable candidate for the study.
14. Patients who have a history of or current diagnosis of glaucoma or posterior subcapsular cataracts or any other ocular condition that, in the opinion of the Investigator, would place study patient at undue risk.
15. Patient is currently receiving or has received any radiation therapy or anti-neoplastic agents within 3 months before baseline.
16. Use within 4 weeks before baseline of 1) oral or intravenous corticosteroids, 2) UVA/UVB therapy, 3) PUVA (psoralen plus ultraviolet A therapy, 4) prescription strength anti-inflammatory agents, 5) topical tacrolimus or pimecrolimus or 6) any other systemic psoriasis treatment.
17. Known history of hypothalamic-pituitary-adrenal axis impairment or any other disturbance of the adrenal function (e.g., Cushing or Addison disease).
18. Use of tanning booths or nonprescription UV light source within 2 weeks before baseline.
19. Use within 8 weeks before baseline of 1) immunomodulators or immunosuppressive therapies, 2) interferon or 3) systemic retinoids.
20. Use within 14 days before baseline of 1) systemic antibiotics, 2) calcipotriene or other Vitamin D preparations, or 3) topical retinoids.
21. Patients who have used topical treatments, prescription or over the counter, including:

    1. Any topical anti-psoriatic therapeutic agents of any kind within the 2 weeks before baseline.
    2. Any topical corticosteroids within the 2 weeks before baseline.
    3. Any antibacterial, medicated and/or astringent washes, soaps, pads or moisturizers within 3 days before baseline.
    4. High strength (20% or above) alpha-hydroxy acid or any kind of peel or other procedures (e.g., laser hair removal) within 30 days before baseline.
    5. Any topical products (i.e., sunscreens, lotions, creams), except for bland emollient (moisturizer) within 24 hours before baseline.
    6. Topical antibiotics in the treatment area within 7 days before baseline.
    7. New regimens of beta blockers.
    8. Lithium preparations within 2 weeks before baseline.
    9. Anti-malarial agents within 2 weeks before baseline.
22. Patient has been treated within 6 months before baseline with any biological therapies for psoriasis.
23. Inability to understand the protocol requirements, instructions, and study related restrictions, the nature, scope, and possible consequences of the clinical study.
24. Unlikely to comply with the protocol requirements, instructions, and study-related restrictions, such as uncooperative attitude, inability to return for follow-up visits, and improbability of completing the clinical study.
25. Receipt of any drug as part of a research study within 30 days before baseline.
26. The patient is a member of the investigational study staff or a member of the family of the investigational study staff.
27. Previous participation in this study.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the IGA score at Day 28 | 28 days
  Patients will be considered to have shown improvement in disease severity if the IGA score decreases by at least one unit from the baseline score, and will be considered a treatment success if the IGA score is either 0 (clear) or 1 (minimal).

SECONDARY OUTCOMES:
Hypothalamic Pituitary Adrenal (HPA) Axis suppression | 28 days
  Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence, defined by 30 minute post- CortrosynTM injection level cortisol level of ≤18 mcg/100 mL, at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rajinder k Jalali, MD, Study Director — Sun Pharmaceutical Industries Limited

IPD SHARING:
Plan to Share IPD: Undecided